CLINICAL TRIAL: NCT05150587
Title: A Phase IIa, Multicenter, Double Blind, Placebo Controlled, Randomized Clinical Trial to Assess Safety, Efficacy and Pharmacokinetics of Rifaximin Delayed-Release (Rifaximin-EIR) in Patients With Moderate-to-severe Papulopustular Rosacea
Brief Title: Safety, Efficacy and Pharmacokinetics of Rifaximin in Patients With Moderate-to-severe Papulopustular Rosacea
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alfasigma S.p.A. (Industry)
Collaborators: bioRASI, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RE-ROS2002-2021
Record Dates: First submitted 2021-10-25; First posted 2021-12-09 (Actual); Results first posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2023-05

CONDITIONS: Papulopustular Rosacea
MeSH Terms: conditions — Rosacea | interventions — Rifaximin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Rifaximin 250 mg TID (Active Comparator)
  Interventions: Drug: Rifaximin
- Rifaximin 500 mg TID (Active Comparator)
  Interventions: Drug: Rifaximin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rifaximin — Rifaximin tablets
  Arms: Rifaximin 250 mg TID; Rifaximin 500 mg TID
Drug: Placebo — Placebo tablets
  Arms: Placebo

SUMMARY:
Rosacea is a common chronic inflammatory relapsing-remitting skin condition almost exclusively affecting the central area of the face and the eyes.

Preliminary evidence suggests that treatment with rifaximin, a poorly absorbed oral antibiotic drug may be beneficial in patients with rosacea, particularly in those with papulopustular phenotype and positivity to Lactulose Breath Test (L-BT).

The objective of this study is twofold:

1. To explore the safety and efficacy of 2 doses of oral Rifaximin versus placebo in adults with moderate-to-severe papulopustular rosacea.
2. To assess the pharmacokinetics (PK) of these two dose regimens in a sub-group of patients.

ELIGIBILITY:
Main Inclusion Criteria:

* Men and women aged 18 years or older at screening.
* Female participants are eligible if they are: i) of non-childbearing potential or ii) of childbearing potential with a negative pregnancy test result at screening and randomization AND agreeing to use a highly effective method of contraception until 72 hours after taking the last study treatment dose.
* Presence of rosacea, papulopustular phenotype.
* Presence of ≥11 and ≤70 facial papules and/or pustules.
* Moderate or severe rosacea based on Investigator's Global Assessment based on Investigator's judgement.
* Patients accepting to provide and legally capable of providing free and informed consent to all procedures included in the protocol (including the availability to perform a Lactulose Breath Test).

Main Exclusion Criteria:

* Granulomatous rosacea or rosacea fulminans.
* Erythematotelangiectatic, phymatous or ocular rosacea only. Patients with these subtypes associated with papulopustular rosacea can be enrolled.
* Rosacea with Investigator's Global Assessment (IGA) grade ≤2 based on Investigator's judgment.
* Anticipated need for proctoscopy or colonoscopy within two weeks after lactulose breath test.
* Subjects requiring a low galactose diet.
* Hypersensitivity or intolerance to lactulose or any excipient of the lactulose reparation to be used for L-BT.
* History of inflammatory bowel disease (Crohn's disease or ulcerative colitis) or other conditions characterized by severe intestinal ulcers.
* History of coeliac disease.
* Patients with intestinal obstruction or partial intestinal obstruction.
* Presence of diarrhoea associated with fever and/or blood in the stool.
* Severe kidney impairment (i.e. estimated glomerular filtration rate <30 ml/min).
* Severe hepatic impairment (i.e. Child-Pugh B or C).
* Cancer or any cancer-related treatment within 5 years prior to screening (excluding non-melanoma skin-cancer).
* History of alcohol or drug abuse within a year prior to screening, based on Investigator's judgement.
* Facial skin conditions that can interfere with reliable assessment of rosacea throughout the study (e.g. facial hair, tattoos, other facial adornments, keloids, hypertrophic scarring, recent facial surgery, excessive sun exposure including use of tanning beds)
* Any other significant health condition (e.g. cardiovascular, respiratory, renal, hepatic, neurologic, psychiatric, hematologic, oncologic, immune etc.) or non-health condition that in the investigator's judgement may: i) jeopardize the patient's safe participation in the trial or ii) make unlikely the patient's completion of the study or iii) make unlikely the patient's compliance with the study procedures (e.g. highly anticipated need of non-permitted treatments, terminal illness, etc.).
* History of hypersensitivity to the study drug.
* Treatment with biologic immunomodulatory and/or immunosuppressive drugs (e.g. anti-tumor necrosis factor [TNF] drugs) within 6 months prior to randomization.
* Treatment with non-biologic immunomodulatory and/or immunosuppressive drugs (e.g. cyclosporine, methotrexate etc.) within 30 days prior to randomization.
* Treatment with warfarin (or other coumarins) within 14 days prior to randomization.
* Treatment with niacin within 30 days prior to randomization.
* Topical facial or systemic antibiotics within 30 days before randomization;
* Treatment with neomycin or other low-absorbable oral antibiotics within 90 days before randomization.
* Topical facial, inhaled or systemic corticosteroids within 30 days prior to randomization.
* Topical facial retinoids within 30 days before randomization.
* Systemic retinoids within 6 months before randomization.
* Any other topical or systemic treatment for rosacea within 30 days before randomization (including also laser and pulsed light, etc.).
* Over-the-counter intestinal or topical skin probiotics (functional food is allowed), within 30 days before randomization.
* Any experimental treatment within 6 months prior to randomization.
* Current swab-positive or suspected (under investigation) Covid-19 infection; or fever and one or more of the following respiratory disease signs or symptoms: cough, sputum production, shortness of breath within the last 14 days; or contact with people with Covid-19 infection within the last 14 days.
* Women who are pregnant, breast-feeding or planning a pregnancy during the trial period.
* Subjects who are investigational site staff members and their family members, site staff members otherwise supervised by the investigator, or patients who are Alfasigma's employees.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2021-10-05 (Actual); Primary Completion 2022-10-20 (Actual); Study Completion 2022-10-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (38):
- United States (38):
  - Dermatology Research Ventures, Yuma, Arizona
  - Johnson Dermatology, Fort Smith, Arkansas
  - Long Beach Clinical Trials, Long Beach, California
  - Metropolis Dermatology, Los Angeles, California
  - LA Universal Research Center, Los Angeles, California
  - Cosmetic Laser Dermatology, San Diego, California
  - UCSD, San Diego, California
  - University Clinical Trials, Inc., San Diego, California
  - Skin Care Research, Boca Raton, Florida
  - MOORE Clinical Research,Inc., Brandon, Florida
  - Sweet Hope Research Specialty, Inc., Hialeah, Florida
  - Savin Medical Group, Miami Lakes, Florida
  - Leavitt Medical Associates of Florida, Ormond Beach, Florida
  - DelRicht Research, Marietta, Georgia
  - DS Research, Clarksville, Indiana
  - Skin Science PLLC, Louisville, Kentucky
  - DS Research, Louisville, Kentucky
  - Delricht Research Baton Rouge LA, Baton Rouge, Louisiana
  - Delricht Research Covington LA, Covington, Louisiana
  - DelRicht Research Houma Louisiana, Houma, Louisiana
  - DelRicht Research, New Orleans, Louisiana
  - Revival Research Institute, LLC., Troy, Michigan
  - Grekin Skin Care Institute, Wyandotte, Michigan
  - MediSearch Clinical Trials, Saint Joseph, Missouri
  - JDR Dermatology Research, Las Vegas, Nevada
  - JUVA Skin and Laser Center, New York, New York
  - Onsite Clinical Solutions, Charlotte, North Carolina
  - Dermatology Consulting Services, PLLC, High Point, North Carolina
  - DelRicht Research, Tulsa, Oklahoma
  - Oregon Dermatology and Research Center, Portland, Oregon
  - Paddington Testing Co, Inc, Philadelphia, Pennsylvania
  - Dermatology Treatment and Research Center, Dallas, Texas
  - 3A Research, El Paso, Texas
  - DelRicht Research Frisco Texas, Frisco, Texas
  - Austin Institute for Clinical Research, Pflugerville, Texas
  - Progressive Clinical Research, San Antonio, Texas
  - Velocity Clinical Research, Salt Lake City, Utah
  - West End Dermatology Associates, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Rifaximin 250 mg TID: 1 tablet of Rifaximin 250 mg TID (750 mg daily) + 1 tablet of placebo TID
- Rifaximin 500 mg TID: 2 tablets of Rifaximin 250 mg formulation TID (1500 mg daily)
- Placebo: 2 tablets of placebo TID
Period: Overall Study
Arm/Group | Rifaximin 250 mg TID | Rifaximin 500 mg TID | Placebo
Started | 70 | 80 | 66
Number of Participants Included in the "Full Analysis Set" | 65 | 76 | 63
Completed | 64 | 73 | 60
Not Completed | 6 | 7 | 6

BASELINE CHARACTERISTICS:
Population: Baseline analysis is based on the Full Analysis Set
Groups:
- Rifaximin 250 mg TID: 1 tablet of Rifaximin 250 TID (750 mg daily) + 1 tablet of placebo TID
- Rifaximin 500 mg TID: 2 tablets of Rifaximin 250 mg TID (1500 mg daily)
- Total: Total of all reporting groups
Arm/Group | Rifaximin 250 mg TID | Rifaximin 500 mg TID | Placebo | Total
Number analyzed (Participants) | 65 | 76 | 63 | 204
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 58 | 67 | 54 | 179
  >=65 years | 7 | 9 | 9 | 25
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 54 | 44 | 150
  Male | 13 | 22 | 19 | 54
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 0 | 2
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1 | 2
  Black or African American | 2 | 4 | 6 | 12
  White | 59 | 68 | 56 | 183
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 3 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Co-primary Endpoint: Change From Baseline in Number of Rosacea Inflammatory Lesions
Description: This is a co-primary endpoint. Success of the study will be declared in any of the active treatment groups if both the co-primary efficacy endpoints (here listed as 1 and 2) will be satisfied (note: the two items may not necessarily occur in the same patient):
  1. Mean change from Baseline in number of rosacea inflammatory lesions (papules, pustules or plaques) at the end of treatment;
  2. Percent of participants showing treatment success defined as IGA (Investigator's Global Assessment) score of 0 or 1 (0=clear; 1=almost clear; 2=mild; 3=moderate; 4=severe) at the end of treatment.
Time Frame: 30 days
Population: The primary efficacy outcomes measures are reported on the Full Analysis Set
Measure: Mean (Standard Deviation); unit: lesions (rosacea inflammatory)
Groups:
- Rifaximin 250 mg TID; Rifaximin 500 mg TID: 2 tablets of Rifaximin 250 mg formulation TID (1500 mg daily)
Arm/Group | Rifaximin 250 mg TID | Rifaximin 500 mg TID | Placebo
Number analyzed (Participants) | 65 | 76 | 63
lesions (rosacea inflammatory) | -10.0 (9.24) | -6.7 (14.78) | -9.2 (10.49)

2. Primary Outcome: Co-primary Endpoint: Treatment Success Rate
Description: as for outcome 1
Time Frame: 30 days
Population: The primary efficacy outcomes measures are reported on the Full Analysis Set
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Rifaximin 250 mg TID | Rifaximin 500 mg TID | Placebo
Number analyzed (Participants) | 65 | 76 | 63
Percentage of participants | 9.23 [2.19 to 16.27] | 9.21 [2.71 to 15.71] | 11.11 [3.35 to 18.87]

ADVERSE EVENTS:
Time Frame: Up to 60 days
Arm/Group | Rifaximin 250 mg TID | Rifaximin 500 mg TID | Placebo
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/80 | 0/66
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/80 | 0/66
Other Adverse Events (participants affected / at risk) | 8/70 | 17/80 | 12/66
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rifaximin 250 mg TID (N=70) | Rifaximin 500 mg TID (N=80) | Placebo (N=66)
headache (Nervous system disorders) | 4 | 4 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 4 | 2
Constipation (Gastrointestinal disorders) | 1 | 3 | 2
Abdominal distension (Gastrointestinal disorders) | 2 | 2 | 1
Nausea (Gastrointestinal disorders) | 1 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 1
Influenza like illness (General disorders) | 0 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-03-25): https://cdn.clinicaltrials.gov/large-docs/87/NCT05150587/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-10): https://cdn.clinicaltrials.gov/large-docs/87/NCT05150587/SAP_001.pdf